CLINICAL TRIAL: NCT06078683
Title: Effects of Acute and Chronic Ketone Ester Consumption on Exercise Tolerance and Cardiac Function in Subjects With the Metabolic Phenotype of Heart Failure With Preserved Ejection Fraction
Brief Title: Effects of Ketone Ester Consumption on Exercise Tolerance and Cardiac Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Yuchi Han, Professor-Clinical, Cardiovascular Medicine, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022H0376; CDMRP-PR212399-F (Other Grant/Funding Number: Departent of Defense)
Record Dates: First submitted 2023-09-26; First posted 2023-10-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Type 2 Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketone Ester (Experimental): This arm will provide a Keto Ester Beverage for consumption.
  Interventions: Dietary Supplement: C8 Ketone Supplement
- Placebo (Placebo Comparator): This arm will provide a Placebo Beverage for consumption.
  Interventions: Dietary Supplement: Placebo
- Keto Ester Acute (Experimental): This arm will provide a Keto Ester Beverage for consumption.
  Interventions: Dietary Supplement: Ketone Ester Acute
- Placebo Acute (Placebo Comparator): This arm will provide a Placebo Beverage for consumption.
  Interventions: Dietary Supplement: Placebo Acute

INTERVENTIONS:
Dietary Supplement: C8 Ketone Supplement — Nutritional and Dietary Manipulation:
  Participants will undertake a controlled feeding intervention where they will drink the supplement twice a day for 6 weeks. The supplement is a C8 Ketone Diester supplement. The beverage contains 25 g of C8 Ketone Diester emulsified in a matrix of water, whey protein concentrate, modified gum acacia, natural and artificial flavors and cocoa powder. It contains 210 kcal, 0.5 g fat, 2 g carbohydrate, and 2 g protein. For the proposed studies all participants will drink 5.4 oz of supplement, delivering 50g of C8 Ketone Supplement daily in a split serving fashion where half will be consumed in the morning with breakfast, and the other half with lunch.
  Arms: Ketone Ester
Dietary Supplement: Placebo — Nutritional and Dietary Manipulation:
  Participants will undertake a controlled feeding intervention where they will drink the placebo twice a day, once at breakfast, and once around lunch time for 6 weeks. The placebo is flavor, energy, volume, and macronutrient matched will be given to patients as part of the placebo arm of the study. This placebo will not contain any ketones (BHB), which will be replaced with a similar caloric content of fat in the form of canola oil.
  Arms: Placebo
Dietary Supplement: Ketone Ester Acute — Nutritional and Dietary Manipulation:
  Participants will undertake a controlled feeding intervention where they will drink two servings of the supplement at once (50g total C8 Ketone Supplement), and images obtained before and after consumption. The supplement is a C8 Ketone Supplement. The beverage contains 25 g of C8 Ketone Diester emulsified in a matrix of water, whey protein concentrate, modified gum acacia, natural and artificial flavors and cocoa powder. It contains 210 kcal, 0.5 g fat, 2 g carbohydrate, and 2 g protein.
  Arms: Keto Ester Acute
Dietary Supplement: Placebo Acute — Participants will undertake a controlled feeding intervention where they will drink two servings of the placebo at once (50g total placebo), and images obtained before and after consumption. The placebo is flavor, energy, volume, and macronutrient matched will be given to patients as part of the placebo arm of the study. This placebo will not contain any BHB, which will be replaced with a similar caloric content of fat in the form of canola oil.
  Arms: Placebo Acute

SUMMARY:
This study is being done to evaluate how a ketone ester (KE) beverage affects heart function and health in people with heart failure compared to a placebo beverage (a beverage made with standard food ingredients that do not contain ketone esters).

DETAILED DESCRIPTION:
This study is a single center, randomized controlled study of up to 30 subjects with metabolic heart failure with preserved ejection fraction (HFpEF) phenotype. The study is designed to compare the effects of KE versus an energy and volume matched placebo on maximal exercise performance measured by CPET. Eligible subjects will have a known diagnosis of HF or type 2 diabetes or metabolic syndrome or obesity and will be selected from a larger population being followed in the Heart Failure Clinic at the Ohio State University Wexner Medical Center. Enrolled subjects will be stratified by sex to ensure equal proportions of men and women in each group (KE and placebo) and then randomly assigned (1:1) to a group, before washing out and crossing over to the other group (KE or Placebo). Subjects will follow the intervention of twice daily consumption of the KE or placebo for a period of 6 weeks, followed by a 4 week washout. All subjects will then crossover to the other group (KE or placebo) for another 6 weeks of intervention. Primary data will be collected at baseline and at the end of the 6-week intervention for both groups. In addition, subjects will undergo daily monitoring of blood markers, blood pressure, heart rate, and overall health. All subjects will continue standard HF and diabetes therapies with adjustment in medications as needed.

Cardiopulmonary exercise testing (CPET) also known as Maximal oxygen consumption testing (VO2) will be used to assess exercise performance, and Cardiac Magnetic Resonance Imaging (CMR) to evaluate cardiac function, myocardial blood flow, and cardiac and vascular function. CMR will provide insightful data on the magnitude, timeline, and functional impact of nutritional ketosis on cardiovascular function in patients diagnosed with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old
2. NYHA class I - III for at least 3 months
3. Ejection fraction ≥ 50% by biplane 2D echo, 3D echo, or CMR.
4. Echo findings of abnormal of indeterminant diastolic function or Right right heart catheterization (RHC) data: At rest: mean pulmonary capillary wedge pressure (PCWP) > 15 mmHg. pulmonary vascular resistance (PVR) < 3 Wood Units
5. Stable medical therapy for at least 3 months as determined by the treating physician (no new cardiac or diabetic medications within 3 months of enrollment, or during enrollment) and dosage should be stable for 1 month prior to enrollment). Dose down titration and discontinuation is allowed during the study
6. Dose of oral diuretics changes allowed, but must be stable for 1 week prior to randomization
7. Body Mass Index (BMI) ≥ 25 and ≤ 50 or Type II Diabetes Mellitus or prediabetes as defined by fasting glucose of 100 - 125 mg/dL or glycated hemoglobin (A1C) 5.7-6.4%, or metabolic syndrome

   a. To meet definition of metabolic syndrome (NCEP ATPIII), 3 of the following criteria must be met: i. Abdominal obesity, defined as a waist circumference ≥102 cm (40 in) in men and ≥88 cm (35 in) in females ii. Serum triglycerides ≥150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides iii. Serum high-density lipoprotein (HDL) cholesterol <40 mg/dL (1 mmol/L) in males and <50 mg/dL (1.3 mmol/L) in females or drug treatment for low HDL cholesterol iv. Blood pressure ≥130/85 mmHg or drug treatment for elevated blood pressure v. Fasting plasma glucose (FPG) ≥100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose
8. Ability to participate in exercise treadmill testing
9. Ability to sign written consent

Exclusion Criteria:

1. Women who are pregnant, current breast-feeding, or have intention to become pregnant while in the trial
2. Known allergy or sensitivity to Gadolinium based contrast agents
3. Implanted pacemaker, cardioverter defibrillator, cardiac resynchronization therapy, left ventricular assist device
4. Other metallic implants/aneurysm clips that are contraindicated in MRI
5. Claustrophobia
6. History of severe kidney disease with estimated glomerular filtration rate (eGFR) <30 ml/kg/1.73m2
7. Type I diabetes
8. History of diabetic ketoacidosis
9. Prescription use of sodium-glucose cotransporter-2 inhibitors (SGLT2i)
10. Prior diagnosis of oxygen dependent pulmonary disease
11. Body Mass Index (BMI) < 25
12. Recent acute myocardial infarction or acute coronary syndrome (30 days)
13. Recent (within 30 days) or planned (within 30 days) cardiac revascularization.
14. History of un-revascularized left main coronary artery disease, severe un- revascularized triple vessel disease, coronary artery bypass graft surgery < 30 days.
15. Left ventricular ejection fraction < 50%
16. Uncontrolled systemic systolic/diastolic blood pressure (SBP/DBP) hypertension (SBP >180 or DBP >110 mmHg)
17. Severe stenotic or regurgitant valvular heart disease, expected to lead to surgery during the trial period.
18. Persistent atrial fibrillation.
19. History of uncontrolled or untreated ventricular arrhythmias
20. Cardiovascular diseases or treatments that increase the unpredictability of the subject's clinical course, independent of heart failure
21. Heart transplant or listing for heart transplant.
22. Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, cardiomyopathy with reversible causes (e.g. stress cardiomyopathy), hypertrophic obstructive cardiomyopathy or known pericardial constriction
23. Acute decompensated heart failure requiring intravenous diuretics, vasodilators, inotropic agents or mechanical support within 1 week of screening and during the screening period prior to randomization
24. Hemoglobin of <9 g/dL at screening
25. Major surgery (major according to the investigator's assessment) performed within 90 days prior to screening, or major scheduled elective surgery (e.g. hip replacement) within 90 days after screening
26. Acute or chronic liver disease, defined by serum levels of transaminases or alkaline phosphatase more than three times the upper limit of normal at screening
27. Gastrointestinal surgery or gastrointestinal disorder that might interfere with supplement consumption. Prior bariatric surgery allowed if weight-stable for past 3 months.
28. Any documented active or suspected malignancy or history of malignancy within 2 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or low-risk prostate cancer (subjects with pre-treatment prostate-specific antigen levels of <10 ng/mL, and biopsy Gleason scores of ≤6 and clinical stage T1c or T2a)
29. Presence of any disease other than heart failure that results in a life expectancy of <1 year (in the opinion of the investigator)
30. History or recurrent severe hypokalemia, potassium < 3.0 mg/dL.
31. Current enrolment in another investigational device or drug study or completion within <30 days of a trial of another investigational device or drug study.
32. Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, will make the subject unlikely to fulfil the trial requirements or complete the trial
33. Any other clinical condition that might jeopardize subject safety during participation in this trial or prevent the subject from adhering to the trial Protocol.
34. Unable or unwilling to follow guidelines of assigned supplement group.
35. Allergy to test article ingredients, or lactose intolerance
36. The subject cannot currently be on a low-carb diet plan. 30-day washout would be required.
37. Patient must have stable weight over the past 3 months (± 5% total body weight). If no weight was recorded in the past 3 months, will have 1 month lead in time for wash out.
38. Refusal to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal exercise performance | Baseline, 6 weeks, 10 weeks, 16 weeks
  Participants will undergo VO2 max testing, conducted by trained professionals. V02 max testing analyses will determine changes in maximal exercise performance

SECONDARY OUTCOMES:
Change in CMR measures of cardiac function | Baseline, 6 weeks, 10 weeks, 16 weeks
  Participants undergo MRI scans, conducted by trained professionals. MRI imaging analyses will determine cardiac function. The images will be analyzed by trained imaging professionals to determine overall change in cardiac function.
Change in New York Heart Association (NYHA) class | Baseline, 6 weeks, 10 weeks, 16 weeks
  NYHA class will be determined by clinical examination by a qualified physician.
Change in Quality of Life Questionnaire | Baseline, 6 weeks, 10 weeks, 16 weeks
  Participants will complete a quality of life questionnaire several times throughout the study. The questions are divided into three areas: Dyspnea, Fatigue and Emotional Function. The scores for each are added up and divided by the number of questions. A 7-point scale is used for areas where 1 is the best and 7 is the worst.
Metabolic Panel | Baseline, 6 weeks, 10 weeks, 16 weeks
  Changes in metabolic blood panel will be assessed at lab visits.
Lipid Panel | Baseline, 6 weeks, 10 weeks, 16 weeks
  Changes in lipid blood panel will be assessed at lab visits.
B-natriuretic peptide (BNP) | Baseline, 6 weeks, 10 weeks, 16 weeks
  Changes in BNP (pg/mL) will be assessed at lab visits.
Change in Cardiac function after acute ingestion of KE or placebo | Baseline, 6 weeks, 10 weeks, 16 weeks
  Cardiovascular performance and function will be investigated using CMR at rest, both before and immediately after consumption of KE or placebo.

OTHER OUTCOMES:
Change in fat storage | Baseline, 6 weeks, 10 weeks, 16 weeks
  Participants undergo Magnetic Resonance Elastography scans, conducted by trained professionals. MRI imaging analyses will determine fat storage.
Change in stiffness | Baseline, 6 weeks, 10 weeks, 16 weeks
  Participants undergo Magnetic Resonance Elastography scans, conducted by trained professionals. MRI imaging analyses will determine stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Han, MD, MMSc, Principal Investigator — Ohio State University
Locations (1):
- The Ross Heart Hospital, Columbus, Ohio, United States